CLINICAL TRIAL: NCT01295086
Title: Dose Determination of Taxotere®, Eloxatin® and Xeloda® (TEX)in Combination With Herceptin® as First-line Treatment for Patients With HER2 Positive Non-resectable Oesophagus, Cardia or Gastric Cancer (ECV)
Brief Title: Taxotere®, Eloxatin® and Xeloda® (TEX) in Combination With Herceptin® as Treatment for HER2 Positive Non-resectable Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Per Pfeiffer, Professor, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Her-TEX
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Adenocarcinoma
Keywords: Adenocarcinoma of the gastro-esophageal; Her2; Dose finding; Taxotere (Docetaxel); Eloxatin (Oxaliplatin); Xeloda (Capecitabine); Herceptin (Trastuzumab)
MeSH Terms: conditions — Adenocarcinoma | interventions — Docetaxel; Oxaliplatin; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Her-TEX (Experimental)
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Docetaxel — 42, 51 or 60 mg/m² day 1 every 3. week
  Other Names: Taxotere
Drug: Oxaliplatin — 100 mg/m² day 1 every 3. week
  Other Names: Eloxatin
Drug: Capecitabine — 1250 mg/² continuously
  Other Names: Xeloda
Drug: Trastuzumab — Trastuzumab 8 mg/kg day 1, cycle 1. Following cycles 6 mg/kg every 3. week
  Other Names: Herceptin

SUMMARY:
The primary aim of this dose-finding study is to determine the maximum tolerated dose of taxotere, eloxatin and capecitabine (TEX) in combination with herceptin given every third week as first-line treatment in patients with HER2-positive advanced gastro-esophageal cancer. Secondary end points are to evaluate progression-free survival and overall survival.

DETAILED DESCRIPTION:
Primary aim:

To define the maximum tolerated dose of the combination of taxotere, eloxatin and capecitabine (TEX) in combination with herceptin given every third week as first- line treatment in patients with HER2-positive advanced gastro-esophageal cancer.

Secondary aims:

Estimating response-rate, progression free survival and overall survival

Methods:

This dose-finding study is planned to include 15 patients with HER2 positive gastro-esophageal cancer, adenocarcinoma. Patients will be included in cohorts of three at progressively higher dose levels.

Chemotherapy will be repeated day 1 every third week to a maximum of eight cycles. Treatment with trastuzumab will continue until disease progression. Dose-limiting toxicity (DLT) will be evaluated after the first cycle. In case of DLT among one of the three patients during the first course of treatment additional three patients will be added at the respective dose level. Dose escalation is continued if 0/3 or 1/6 patients experience DLT.

Patients will be evaluated with a ct- scan at baseline and after every three cycles to exclude progression and evaluate response. Response is assessed by investigators according to RECIST version 1.1.

Blood counts regarding tumour biology will be collected at baseline before 2nd, 4th and 7th cycle and 4 weeks after ended treatment. After completion of treatment patients will be followed every third month until progression or death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven ECV-adenocarcinoma, non-resectable or metastatic disease
2. HER2-positive tumor tissue (IHC 3 + or FISH positive)
3. LVEF > 50 % (MUGA scan or echocardiography)
4. Age ≥ 18 years
5. No prior chemotherapy
6. WHO performance status 0-1
7. Life expectancy of at least 3 months
8. Neutrophils ≥ 1.5 x 109/L and platelets ≥ 100 x 109/L
9. Bilirubin ≤ 1.5 x UNL (Upper Normal Limit) and ASAT and/or ALAT ≤ 3 x UNL. In case of liver metastases no UNL for ASAT and ALAT
10. Creatinine clearance ≥ 50 ml/min. Calculated with the Cockroft-Gault formula
11. No neuropathy
12. Planned treatment start within 8 days after inclusion

Exclusion Criteria:

1. Patients who cannot complete treatment or evaluation
2. Any condition or treatment which after the opinion of the investigator may expose the patients to a risc or influence the purpose of the study
3. Known hypersensitivity towards any of the study drugs
4. Other malignant disease within the last 5 days, except for non-melanoma skin cancer
5. Other serious disease (e.g. cardiac disease, AMI within 1 year or infection)
6. Pregnant women or nursing women
7. Physical or mental conditions which may prevent absorption of oral treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
To determine maximum tolerable dose (MTD) for the combination regime TEX | 2 years
  The investigators have planned to examine 3 dose levels including 3 patients at each level with escalating doses of docetaxel from 42 mg/m² to 60 mg/m² and fixed doses of oxaliplatin (100 mg/m²), capecitabine 625 mg/m² x 2 and trastuzumab 6 mg/kg.

SECONDARY OUTCOMES:
Progression free survival | 3 years
  Time from inclusion to disease progression or death of any cause.
Survival | 4 years
  Time from inclusion to death of any cause.
Response rate | 3 years
  According to RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, Professor, Study Chair — Odense University Hospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense